CLINICAL TRIAL: NCT05690321
Title: Opium Tincture Against Chronic Diarrhea - Patients An Investigator Initiated, Randomized Placebo-controlled, Double-blinded, Clinical Trial
Brief Title: Opium Tincture Against Chronic Diarrhea - Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asbjørn Mohr Drewes (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Asbjørn Mohr Drewes, Professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dropizol_patients; 2020-000396-20 (EudraCT Number)
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Chronic Diarrhea
Keywords: Diarrhea; Gastrointestinal transit
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator): Administration of opium tincture (Dropizol)
  Interventions: Drug: Opium tincture
- Placebo treatment (Placebo Comparator): Administration of placebo (identical to opium tincture in taste and appearance)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Opium tincture — Self-administration of opium tincture (10 mg/ml) as 3x5 drops on day 1-3, 3x10 drops on days 4-6, and 1x10 drops on day 7 in each study period
  Other Names: Dropizol
  Arms: Active treatment
Drug: Placebo — Self-administration of placebo (10 mg/ml) as 3x5 drops on day 1-3, 3x10 drops on days 4-6, and 1x10 drops on day 7 in each study period
  Arms: Placebo treatment

SUMMARY:
The purpose of this study is to investigate the mechanistic anti-propulsive effects of opium tincture on the gastrointestinal tract of a cohort of patients with chronic diarrhea

DETAILED DESCRIPTION:
Opium tincture is used a symptomatic drug against chronic diarrhea even though no clinical studies have investigated the effect on gastrointestinal function. With this randomized, double-blind, placebo-controlled cross-over trial in 16 patients with chronic diarrhea, we wish to provide evidence-based insights into the effects of opium tincture on gastrointestinal function. Additionally, effects on the central nervous system will be investigated a tertiary aim.

ELIGIBILITY:
Inclusion Criteria:

* • Signed informed consent before any study specific procedures

  * Able to read and understand Danish
  * Male or female with an age of 20 years or more
  * The researcher believes that the participant understands what the study entails, are capable of following instructions, can attend when needed, and are expected to complete the study.
  * The investigator will ensure that fertile female participants have a negative pregnancy test before each treatment visit and use contraception during the entity of the study.
  * Specific underlying pathophysiology has been identified, but targeted treatment (e.g. antibiotics or bile acid sequestrants) and treatment with loperamide has failed.

OR

* No specific underlying pathophysiology has been identified and treatment with loperamide has failed.
* At least 6 months post-surgery in the gastrointestinal tract
* No sign of cancer at standard clinical follow-up
* Chronic diarrhea defined as at least 3 daily bowel movements for the last week

Exclusion Criteria:

* • Known allergy towards pharmaceutical compounds similar to Dropizol.

  * Participation in other studies within 14 days of first visit (1 year if opioids involved).
  * Expected need of medical/surgical treatment during the study
  * History of psychiatric illness (e.g. mental retardation, schizophrenia, major depression)
  * History of substance abuse (e.g. alcohol, THC, benzodiazepine, central stimulants and/or opioids)
  * Family history of substance abuse
  * Known major stenosis of the intestines
  * Known severe decreased renal function (defined as eGFR below 30)
  * Known severe decreased hepatic function (defined as Child-Pugh class B or higher)
  * Treatment with MAO- inhibitors during the entity of the study
  * Severe COPD or acute severe asthma (defined as FEV1 below 50 % or acute ongoing exacerbation)
  * Known cor pulmonale
  * Female participants that are lactating
  * Medicine known to affect gastrointestinal motility must not be initiated during the entity of the study
  * Treatment with opium tincture during the last month

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Bowel movement frequency | From day 1 to 7
  Difference in number of spontaneous bowel movements per day between arms

SECONDARY OUTCOMES:
Gastrointestinal transit | Measurement started on day 4 of each study period until expulsion of the capsule]
  Difference in hours from ingestion of a wireless motility capsule to expulsion of the capsule during active and placebo treatment
Stool consistency | From day 1 to 7 in each study period
  Rated on the Bristol Stool Form Scale (ranging from type 1 - type 7)
Pupil diameter | Day 1, 4 and 7 in each study period
  Measured in mm
General cognition | Day 1, 4 and 7 in each study period
  Evaluated using the Mini-Mental State Examination
Reaction time | Day 1, 4 and 7 in each study period
  Measured in milliseconds (ms) from a sound was provided and until the participant pressed a button
Short-term memory | Day 1, 4 and 7 in each study period
  Measured as number of digits correctly remembered after visual presentation
Gastrointestinal symptoms | Day 1, 4 and 7 in each study period
  Measured on the Gastrointestinal Symptom Rating Score (GSRS) questionnaire
Constipation symptoms | Day 1, 4 and 7 in each study period
  Measured on the Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Mohr Drewes, Principal Investigator — Aalborg University Hospital
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Aarhus University hospital, Aarhus

IPD SHARING:
Plan to Share IPD: Yes
Data can by provided upon request
Access Criteria: Researchers who provide a methodological sound proposal

REFERENCES:
- [Derived] Okdahl T, Hoyer KL, Knoph CS, Davidsen L, Larsen IM, Mark EB, Hvas CL, Krogh K, Drewes AM. Opium tincture has anti-propulsive effects in patients with chronic diarrhea: a randomized, placebo-controlled, and cross-over trial. Scand J Gastroenterol. 2024 Sep;59(9):1023-1034. doi: 10.1080/00365521.2024.2381694. Epub 2024 Jul 25. PMID 39054596